CLINICAL TRIAL: NCT00655993
Title: Effect of Statin Therapy on C-reactive Protein Levels in Patients With COPD
Brief Title: Effect of Statin Therapy on C-reactive Protein Levels in Patients With Chronic Obstructive Lung Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Loma Linda Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, James D. Anholm, M.D., Principal Investigator, VA Loma Linda Health Care System
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00746
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: COPD; Inflammation
Keywords: COPD; Inflammation; CRP levels; simvastatin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo drug
  Interventions: Drug: simvastatin
- 2 (Active Comparator): simvastatin
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — 40 mg po daily

SUMMARY:
Hypothesis for this pilot study is that simvastatin will lower the levels of CRP and ET-1 in COPD patients.

DETAILED DESCRIPTION:
Patients with chronic obstructive lung disease (COPD) have an ongoing systemic inflammation, which can be assessed by measuring C-reactive protein (CRP). CRP is found to be a strong and independent predictor of future COPD outcomes. Statins are a class of cholesterol lowering drugs that decrease mortality from cardiovascular disease and stroke. In addition, they have anti-inflammatory, anti-thrombotic and immunomodulatory properties. Statins lower C-reactive protein by the ability to reduce the production of interleukin (IL)-6, the cytokine that activates the acute phase CRP response.

Thus the rationale for this study is to evaluate effect of statins on the levels of CRP and ET-1 in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Medically optimized COPD patients
* Age 40-79 years.
* serum CRP levels >3mg/l

Exclusion Criteria:

* Current smoker
* COPD exacerbation in the last 2 months.
* Active hepatic or severe renal dysfunction.
* connective tissue disease, chronic inflammatory disease, malignancy, any acute illness, leukocytosis (>10,000 white blood cells) or thrombocytosis (>450,000 platelets).
* Recent h/o myocardial infarction, angina in the last 6 months.
* Pregnancy.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
serum CRP levels | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lennard Specht, M.D., Principal Investigator — VA Loma Linda Health Care System; Hemal J. Parekh, M.D., Principal Investigator — VA Loma LInda Healthcare System; James D. Anholm, M.D., Principal Investigator — VA Loma Linda Healthcare System
Locations (1):
- VA Loma Linda Health Care System, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No